CLINICAL TRIAL: NCT06604780
Title: Implementation and Evaluation of a Transition to Discharge Program for the Reduction of Early Readmission in a Mental Health Inpatient Unit
Brief Title: Reducing Early Readmission to an Acute Psychiatric Unit
Acronym: PPREINGRESOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PPREINGRESOTEMP
Record Dates: First submitted 2024-08-14; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-04

CONDITIONS: Readmission; Mental Health Disorder; Hospitalizations Psychiatric
Keywords: early readmission; discharge interventions; psychyatric unit; continuity of care; psychotherapy group; recovery
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group (Experimental): The intervention program is based on the Discharge Transition Model for the prevention of hospital readmission in Mental Health. This is a multicomponent program that initially involves the development of a scale to assess the risk of readmission for each patient, followed by its systematic application. This allows for stratification of patients according to their risk of early readmission and adaptation of the intervention to the needs of each risk level. The intervention includes elements aimed at promoting continuity of care after discharge, transitioning back to the community setting, as well as elements aimed at enhancing personal and emotional resources through psychotherapeutic approaches.
  Interventions: Behavioral: Transitional discharge program
- Control group I (No Intervention): To assess the effectiveness of the Multicomponent Discharge Transition Program, users from Málaga East Axarquía Hospital and North Málaga Health Management Area will be employed as the control group. Participants in the control group will continue with their usual treatment.
- Control group II (No Intervention): Additionally, users from the Mental Health Management Unit of Regional Hospital of Málaga who were admitted the previous year and thus did not participate in the intervention program will also be used as a control group.

INTERVENTIONS:
Behavioral: Transitional discharge program — For patients classified in the low-risk group, general measures would be applied. For patients in the medium-risk group, reinforced measures would be implemented. Lastly, for patients considered to be in the high-risk group, intensive case management measures would be applied, and if they meet the inclusion criteria, they would be included in the Post-Discharge Group Psychotherapeutic Intervention.
  1. General measures
  2. Reinforcement measures
  3. Intensive measures
     * Intensive case management measures
     * Post-Discharge Psychotherapeutic Recovery Support Program: For application to patients at high risk of early readmission who meet the inclusion criteria. It consists of a multicomponent group psychotherapeutic intervention from a rehabilitative and recovery-oriented perspective. This intervention will be structured into 20 sessions, each lasting 90 minutes, held weekly in an open format.
  Arms: Intervention group

SUMMARY:
Early readmission to psychiatric units poses a significant challenge for both patients with mental health issues and healthcare institutions. It hampers patient progress and prognosis, and the professional approach taken during discharge can greatly influence the recovery process. This paper proposes a multicomponent discharge transition intervention to mitigate the risk of early readmission to a Mental Health Hospitalization Unit (MHHU).

The intervention entails developing a measurement scale to assess patients' risk of early readmission, allowing for stratification into high, medium, and low-risk categories. Tailored intervention strategies will focus on ensuring adherence and continuity of care post-discharge, with a more comprehensive approach for high-risk patients. Additionally, a post-discharge psychotherapeutic group will be incorporated for high-risk cases to support recovery. The efficacy of the program will be analyzed by comparing the overall early readmission risk at the Regional Hospital of Malaga's MHHU with the previous year, using admission episodes from two other hospitals in the province as a control group where the intervention program is not implemented. The success of the post-discharge group psychotherapeutic intervention will be evaluated through pre-post assessments of recovery measures, functionality, subjective well-being, social support, and treatment satisfaction.

This proposal aims to address the issue of early readmission to psychiatric units by enhancing predictability and understanding of intervention strategies to reduce readmission rates.

DETAILED DESCRIPTION:
The aim of this study is, firstly, to create a tool for assessing the risk of early readmission that allows for stratification of admitted patients according to their risk level, based on the analysis of clinical and sociodemographic variables. The second objective is to implement an intervention program tailored to each risk level, involving coordination among all involved mental health units and a specific intensive program for patients at higher risk.

The present study is a quasi-experimental cluster clinical trial aimed at assessing the efficacy of a multicomponent discharge transition program for the reduction of early readmissions in a MHHU. The development of this study consists of two distinct parts or elements:

To carry out the main objective, a quasi-experimental design with a control group will be used, and within the intervention, an early readmission risk assessment scale will be created to categorize patients into different risk levels.

In addition, a study will be conducted to assess the predictive value and validity of the early readmission risk rating scale and to study the risk factors for early readmission.

ELIGIBILITY:
Inclusion Criteria:

* All hospital admission episodes at MHHU during the 12 months following the implementation of the Discharge Transition Intervention Program will be considered.
* The experimental group, to which the Discharge Transition Intervention Program will be applied, will consist of users whose Community Mental Health Units (CMHU) are affiliated with the Regional Hospital of Málaga.

Exclusion Criteria:

• Users belonging to other hospitals in the province will be excluded from the intervention program and will form part of the control group.

Post-Discharge Group Psychotherapy Support Recovery has its own eligibility criteria:

Inclusion criteria:

* Be of legal age.
* Speak spanish fluently.
* Have had recent admission to the MHHU of the Regional Hospital of Málaga and a score considered as "High Risk" on the Early Rehospitalization Risk Scale or have experienced an early rehospitalization.
* Belong to the Clinical Management Unit of Mental Health of the RUH of Málaga.
* Have sufficient cognitive capacity to understand the rules and contents of the group intervention.

Exclusion criteria:

* Individuals whose primary diagnosis is a Mental and Behavioral Disorder due to psychoactive substance use.
* Moderate or severe intellectual disability.
* Clinical Management Unit belonging to a hospital other than the RUH of Málaga.
* Lack of commitment to attending sessions or complying with group rules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 836 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Early readmission rate | Data will be collected over the 12 months following the implementation of the intervention program.
  Changes in the percentage of early readmissions over the total number of recorded admission episodes, considering early readmission as any admission episode that occurs within 30 days after hospital discharge.

SECONDARY OUTCOMES:
Recovery | Five months between pre and post evaluation
  Changes in measures of recovery, will be assessed through pre-post administration of the QPR-15-SP questionnaire.
Functionality | Five months between pre and post evaluation
  Changes in measures of functionality, will be assessed through pre-post administration of the PSP questionnaire.
Subjective well-being | Five months between pre and post evaluation
  Changes in measures of subjective well-being, will be assessed through pre-post administration of the Core-Om questionnaire.
Satisfaction with treatment | Five months between pre and post evaluation
  Changes in measures of satisfaction with treatment, will be assessed through pre-post administration of the CAT questionnaire.
Perceived social support | Five months between pre and post evaluation
  Changes in Perceived social support will be assessed through pre-post administration of the DUKE-UNK questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Vera Carbonell Aranda, Bachelor, Principal Investigator — Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud
Locations (1):
- Vera Carbonell Aranda, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tyler N, Wright N, Waring J. Interventions to improve discharge from acute adult mental health inpatient care to the community: systematic review and narrative synthesis. BMC Health Serv Res. 2019 Nov 25;19(1):883. doi: 10.1186/s12913-019-4658-0. PMID 31760955
- [Background] Donisi V, Tedeschi F, Salazzari D, Amaddeo F. Pre- and post-discharge factors influencing early readmission to acute psychiatric wards: implications for quality-of-care indicators in psychiatry. Gen Hosp Psychiatry. 2016 Mar-Apr;39:53-8. doi: 10.1016/j.genhosppsych.2015.10.009. Epub 2015 Nov 1. PMID 26804775
- [Background] Wobrock T, Weinmann S, Falkai P, Gaebel W. Quality assurance in psychiatry: quality indicators and guideline implementation. Eur Arch Psychiatry Clin Neurosci. 2009 Nov;259 Suppl 2(Suppl 2):S219-26. doi: 10.1007/s00406-009-0072-7. PMID 19876682
- [Background] Vigod SN, Kurdyak PA, Seitz D, Herrmann N, Fung K, Lin E, Perlman C, Taylor VH, Rochon PA, Gruneir A. READMIT: a clinical risk index to predict 30-day readmission after discharge from acute psychiatric units. J Psychiatr Res. 2015 Feb;61:205-13. doi: 10.1016/j.jpsychires.2014.12.003. Epub 2014 Dec 13. PMID 25537450
- [Background] Vigod SN, Kurdyak PA, Dennis CL, Leszcz T, Taylor VH, Blumberger DM, Seitz DP. Transitional interventions to reduce early psychiatric readmissions in adults: systematic review. Br J Psychiatry. 2013 Mar;202(3):187-94. doi: 10.1192/bjp.bp.112.115030. PMID 23457182
- [Background] Owusu E, Oluwasina F, Nkire N, Lawal MA, Agyapong VIO. Readmission of Patients to Acute Psychiatric Hospitals: Influential Factors and Interventions to Reduce Psychiatric Readmission Rates. Healthcare (Basel). 2022 Sep 19;10(9):1808. doi: 10.3390/healthcare10091808. PMID 36141418
- [Background] Hegedus A, Kozel B, Richter D, Behrens J. Effectiveness of Transitional Interventions in Improving Patient Outcomes and Service Use After Discharge From Psychiatric Inpatient Care: A Systematic Review and Meta-Analysis. Front Psychiatry. 2020 Jan 21;10:969. doi: 10.3389/fpsyt.2019.00969. eCollection 2019. PMID 32038320
- [Background] García-Herrera Pérez-Bryan JM, Hurtado Lara MM, Quemada González C, Nogueras Morillas EV, Bordallo Aragón A, Martí García C, et al. Guía de Práctica Clínica para el Tratamiento de la Psicosis y la Esquizofrenia. Manejo en Atención Primaria y en Salud Mental. [Internet]. Plan Integral de Salud Mental. Servicio Andaluz de Salud, editor. 2019 [cited 2024 Jan 29]. Available from: https://www.sspa.juntadeandalucia.es/servicioandaluzdesalud/sites/default/files/sincfiles/wsas-media-pdf_publicacion/2020/1gpc_psicosis_completa.pdf
- [Background] Ministerio de Ciencia e Innovación. Guía de Práctica Clínica de intervenciones psicosociales en el trastorno mental grave [Internet]. 2009 [cited 2024 Jan 29]. Available from: https://portal.guiasalud.es/wp-content/uploads/2018/12/GPC_453_TMG_ICS_compl.pdf
- [Background] Lam M, Li L, Anderson KK, Shariff SZ, Forchuk C. Evaluation of the transitional discharge model on use of psychiatric health services: An interrupted time series analysis. J Psychiatr Ment Health Nurs. 2020 Apr;27(2):172-184. doi: 10.1111/jpm.12562. Epub 2019 Sep 29. PMID 31529589
- [Background] Chris Evans JMCFMMBKAJCGM. CORE: Clinical Outcomes in Routine Evaluation. http://dx.doi.org/101080/jmh93247255. 2009 Jan;9(3):247-55.
- [Background] Feixas i Viaplana G, Evans C, Trujillo A, Saúl Gutiérrez LÁ, Botella L, Corbella S, et al. La versión española del CORE-OM: Clinical Outcomes in Routine Evaluation - Outcome Measure. Revista de Psicoterapia. 2012;23(89):109-35.
- [Background] Bellon Saameno JA, Delgado Sanchez A, Luna del Castillo JD, Lardelli Claret P. [Validity and reliability of the Duke-UNC-11 questionnaire of functional social support]. Aten Primaria. 1996 Sep 15;18(4):153-6, 158-63. Spanish. PMID 8962994
- [Background] Broadhead WE, Gehlbach SH, de Gruy FV, Kaplan BH. The Duke-UNC Functional Social Support Questionnaire. Measurement of social support in family medicine patients. Med Care. 1988 Jul;26(7):709-23. doi: 10.1097/00005650-198807000-00006. PMID 3393031
- [Background] Morosini PL, Magliano L, Brambilla L, Ugolini S, Pioli R. Development, reliability and acceptability of a new version of the DSM-IV Social and Occupational Functioning Assessment Scale (SOFAS) to assess routine social functioning. Acta Psychiatr Scand. 2000 Apr;101(4):323-9. PMID 10782554
- [Background] Garcia-Portilla MP, Saiz PA, Bousono M, Bascaran MT, Guzman-Quilo C, Bobes J; en nombre del grupo de validacion de la version espanola de la escala de Funcionamiento Personal y Social (PSP). Validation of the Spanish Personal and Social Performance scale (PSP) in outpatients with stable and unstable schizophrenia. Rev Psiquiatr Salud Ment. 2011 Jan;4(1):9-18. doi: 10.1016/j.rpsm.2010.11.003. Epub 2011 Mar 10. English, Spanish. PMID 23446097
- [Background] Law H, Neil ST, Dunn G, Morrison AP. Psychometric properties of the questionnaire about the process of recovery (QPR). Schizophr Res. 2014 Jul;156(2-3):184-9. doi: 10.1016/j.schres.2014.04.011. Epub 2014 May 9. PMID 24816049
- [Background] Goodman-Casanova JM, Cuesta-Lozano D, Alupoaei C, Grasa Bello EM, Herrera-Imbroda J, Mayoral-Cleries F, Guzman-Parra J. Psychometric validation of the 15-item Questionnaire about the Process of Recovery in Spain (QPR-15-SP). Front Psychol. 2023 Jul 5;14:1178341. doi: 10.3389/fpsyg.2023.1178341. eCollection 2023. PMID 37484089
- [Background] Richardson M, Katsakou C, Torres-Gonzalez F, Onchev G, Kallert T, Priebe S. Factorial validity and measurement equivalence of the Client Assessment of Treatment Scale for psychiatric inpatient care - a study in three European countries. Psychiatry Res. 2011 Jun 30;188(1):156-60. doi: 10.1016/j.psychres.2011.01.020. Epub 2011 Feb 22. PMID 21342706
- [Background] Priebe S, Gruyters T, Heinze M, Hoffmann C, Jakel A. [Subjective evaluation criteria in psychiatric care--methods of assessment for research and general practice]. Psychiatr Prax. 1995 Jul;22(4):140-4. German. PMID 7675903
- [Background] Glenn D, Golinelli D, Rose RD, Roy-Byrne P, Stein MB, Sullivan G, Bystritksy A, Sherbourne C, Craske MG. Who gets the most out of cognitive behavioral therapy for anxiety disorders? The role of treatment dose and patient engagement. J Consult Clin Psychol. 2013 Aug;81(4):639-649. doi: 10.1037/a0033403. Epub 2013 Jun 10. PMID 23750465
- [Background] Spinner EN, Stapleton M, Oppenlander JE, Murray E, Shaikh R, Ramkirpaul E. Utility of the READMIT Index to Identify Community Hospital 30-Day Psychiatric Readmissions. Issues Ment Health Nurs. 2021 Apr;42(4):391-400. doi: 10.1080/01612840.2020.1814910. Epub 2020 Oct 7. PMID 33027602
- [Background] Herrera-Imbroda J. Reingreso psiquiátrico y calidad asistencial. Boletín Psicoevidencias. 2023;65.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT06604780/Prot_SAP_000.pdf